CLINICAL TRIAL: NCT06026826
Title: Intervention Effect of Transcranial Alternating Current Stimulation(tACS) on Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tACS-anxiety
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Transcranial Alternating Current Stimulation; Anxiety Disorder; Magnetic Resonance Imaging
Keywords: Transcranial Alternating Current Stimulation; Anxiety Disorder; Magnetic Resonance Imaging
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active tACS twice daily for one week. The anode was placed over AF3 with return electrodes placed at the contralateral mastoid process. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes per session, twice daily over 7 consecutive days, and the stimulus frequency was set as 8 Hz.
  Interventions: Device: transcranial alternating current stimulation
- sham stimulation (Sham Comparator): Participants will receive sham tACS twice daily for one week. Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: sham transcranial alternating current stimulation

INTERVENTIONS:
Device: transcranial alternating current stimulation — tACS is described as a non-invasive form of brain stimulation that uses a low-intensity, alternating current applied directly to the head through scalp electrodes.
  Arms: real stimulation
Device: sham transcranial alternating current stimulation — Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of transcranial alternating current stimulation(tACS) on anxiety symptoms and somatic symptoms in patients with anxiety disorder and its underlying neural mechanism by MRI.

DETAILED DESCRIPTION:
Forty patients with anxiety disorder diagnosed by DSM-5 were recruited from the second affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving tACS. After meeting the inclusion criteria and obtaining informed consent, each participant will complete the clinical evaluation, functional magnetic resonance imaging (fMRI) and tACS treatment conducted by trained researchers at the Neuropsychological Synergetic Innovation Center of Anhui Medical University. All the participants were randomized (1:1) to receive "active" or "sham" treatment protocol. The anode was placed over AF3 with return electrodes placed at the contralateral mastoid process. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes per session, twice daily over 7 consecutive days, and the stimulus frequency was set as 8 Hz. Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.

Before and after the tACS treatment, the patients had receiving a battery measure of neuropsychological tests and Magnetic resonance imaging scan in multimodalities. Neuropsychological assessment included HAMD, HAMA, PHQ15, ISI, ASI, SAS, RRS, IUS. Multimodal fMRI includes 3D-T1, rs-fMRI and DTI.

Neuropsychological evaluation and magnetic resonance imaging data were obtained again 24 hours after the last treatment. The symptoms of the patients were followed up one month after the end of treatment.They were instructed to focus their answers on the past week. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for anxiety, and HAMA>14, PHQ-15>5.

the age ranged from 18 to 60 years old, and the length of education was more than 5 years.

the visual acuity or corrected visual acuity is normal, right-handed, can cooperate with the completion of various experimental tests.

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.

accompanied by other neurological diseases, such as stroke, epilepsy and so on. pregnant and lactating women. accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective disorder, hysteria, autism and so on.

patients with MRI taboos or factors affecting imaging quality, such as cardiac pacemaker, cochlear implant, cardio-cerebrovascular metal stent, metal denture, etc.

those who could not cooperate with those who completed the relevant experiments, such as patients with depressive stupor, claustrophobia and so on.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
anxiety symptoms | baseline and immediately after intervention
  the change of anxiety symptoms assessed by HAMA scale(Hamilton Anxiety Scale) will constitute the major research outcome measure, to assess response to tACS. HAMA scale scores range from 0 to 56 points, the higher the score indicates the more serious anxiety symptoms
resting-state functional connectivity | baseline and immediately after intervention
  the change of resting-state functional connectivity strength between stimulated target and the whole brain areas will be measured by functional MRI.

SECONDARY OUTCOMES:
somatic symptoms | baseline and immediately after intervention
  the change of somatic symptoms will be assessed by Patient Health Questionnaire (PHQ-15). PHQ-15 is composed of 15 physical symptoms that have been extracted from the PHQ. PHQ-15 scale scores range from 0 to 30 points. Higher scores indicate more severe somatic symptoms.
SAS(Self-rating anxiety scale) | baseline and immediately after intervention
  Self-rating anxiety scale(SAS) is a supplementary evaluation of the change of anxiety state of patients in this experiment, and it also belongs to the category of self-rating scale. Patients assessed anxiety by checking the frequency of 20 items: none or almost none, sometimes, most of the time, most of the time, or all of the time. SAS scale scores range from 0 to 100 points。The higher the score, the more serious the anxiety symptoms.
ISI(The insomnia severity index) | baseline and immediately after intervention
  ISI(The insomnia severity index) is used to evaluate the changes of sleep status of anxiety patients in the recent (2 weeks), which is a self-rating scale. ISI scale scores range from 0 to 28 points. The higher the score is, the worse the sleep quality is. This scale indirectly reflects the changes of patients' anxiety state through evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, China